CLINICAL TRIAL: NCT01719250
Title: A Pilot Study of the PI3K Inhibitor BKM120 in Patients With Relapsed Lymphoma
Brief Title: Buparlisib in Treating Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1183; NCI-2012-01582 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1183 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma; Transformed Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (buparlisib) (Experimental): Patients receive buparlisib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Buparlisib — Given PO
  Other Names: BKM120; PI3K Inhibitor BKM120
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well buparlisib works in treating patients with non-Hodgkin lymphoma that has returned after a period of improvement or has not responded to previous treatment. Buparlisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical benefit rate (complete response [CR], partial response [PR] or standard disease [SD] >= 6 months) with BKM120 (buparlisib) in patients with relapsed or refractory lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate overall response rate, overall survival, progression-free survival and duration of response.

II. To describe the toxicities associated with BKM120 in lymphoma. III. To evaluate prognostic factors for aggressive lymphoma and whether there's a correlation with clinical benefit.

TERTIARY OBJECTIVES:

I. To assess serum cytokines before and after BKM120 therapy. II. To assess phosphatidylinositol 3-kinase (PI3K) pathway member expression on paraffin-embedded tumor samples pre-treatment.

III. To assess on paired fresh tumor tissue obtained from consenting patients pre- and post-therapy the change in activation of PI3K pathway members.

OUTLINE: Patients receive buparlisib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven relapsed, refractory or residual aggressive B-cell non-Hodgkin lymphoma; NOTE: re-biopsy is necessary unless the patient has had a previous biopsy < 168 days prior to registration on this protocol and there has been no intervening treatment; eligible tumor types are diffuse large B-cell non-Hodgkin lymphoma (NHL), mantle cell lymphoma, transformed NHL, and follicular grade III
* Not a candidate or has declined standard salvage therapy for their disease
* Measurable disease as defined by at least ONE of the following:

  * Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) or the CT portion of the positron emission tomography (PET)/CT: must have at least one lesion that has a single diameter of >= 2 cm or tumor cells in the blood >= 5 x 10^9/L
  * Skin lesions can be used if the area is >= 2 cm in at least one diameter and photographed with a ruler
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1000/uL
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets (PLT) >= 100,000/uL
* Serum bilirubin within normal range (or =< 1.5 x upper limit of normal [ULN] if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert syndrome)
* Aspartate aminotransferase (AST) within normal limits or =< 3 x ULN if due to lymphoma
* Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 mL/min
* Magnesium >= lower limit of normal (LLN)
* Potassium >= LLN
* Serum amylase =< ULN
* Serum lipase =< ULN
* Fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
* Serum calcium =< 10.9 mg/dL
* Negative pregnancy test done =< 72 hours prior to starting drug, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Mayo Clinic Rochester for follow-up
* Willing to provide blood samples for correlative research purposes
* Willingness to take BKM120 orally

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ highly effective contraception during dosing with BKM120 and for 4 weeks after the final dose of treatment; NOTE: women of childbearing potential are defined as all women physiologically capable of becoming pregnant
  * Men of childbearing potential who are unwilling to employ highly effective contraception during dosing with BKM120 and for 16 weeks after the final dose of treatment and should not a father a child during this time; NOTE: men of childbearing potential are defined as all males physiologically capable of conceiving offspring

    * NOTE: the highly effective contraception is defined as either:

      * True abstinence: when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
      * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
      * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); for female subjects on the study, the vasectomized male partner should be the sole partner for that patient
      * Use of a combination of any two of the following (a+b):

        1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
        2. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
      * Oral contraception, injected or implanted hormonal methods are not allowed
* Uncontrolled infection
* Average baseline of >= 4 stools per day
* Therapy with myelosuppressive chemotherapy or biologic therapy < 21 days prior to registration unless the patient has recovered from the nadir of the previous treatment to a level that meets the inclusion eligibility criteria of this protocol
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half-lives prior to registration or who have not recovered from side effects of such therapy
* Received wide field radiotherapy =< 28 days or limited field radiation for palliation =< 14 days prior to registration or who have not recovered from side effects of such therapy
* Receiving corticosteroids > 10 mg of prednisone per day (or equivalent); NOTE: patients may be receiving stable doses of corticosteroids with a maximum dose of 10 mg of prednisone per day if they are being given for disorders other than lymphoma such as rheumatoid arthritis, polymyalgia rheumatica or adrenal insufficiency, or asthma
* Persistent toxicities >= grade 2 from prior chemotherapy or biological therapy regardless of interval since last treatment
* Active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 45% as determined by multi gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Fridericia's corrected QT interval (QTcF) > 450 msec on screening electrocardiogram (ECG) (using the QTcF formula)
  * Unstable angina pectoris; patients with unstable angina should have angina controlled before entering the study
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Symptomatic pericarditis
  * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Known positivity for human immunodeficiency virus (HIV); note: baseline testing for HIV is not required
* Active hepatitis B or C with uncontrolled disease; note: a detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) ribonucleic acid (RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior hepatitis B virus (HBV) infection
* Other active malignancy requiring treatment that would interfere with the assessments of response of the lymphoma to protocol treatment
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Any severe and/or uncontrolled medical conditions such as diabetes, poor lung function, or other conditions that, in the treating physician's opinion, could adversely impact their ability to participate in the study
* Patients who have received prior treatment with a P13K inhibitor; patients with prior mammalian target of rapamycin (mTOR) inhibitor therapy are eligible
* Using medications that have a strong risk of prolonging the QT interval or inducing torsades de pointes
* Major surgery =< 14 days prior to registration or have not recovered from side effects of such therapy
* Currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5), (please note that co-treatment with weak inhibitors of cytochrome P450, family 3, subfamily A [CYP3A] is allowed)
* Receiving certain fruits or herbal preparations/medications including, but are not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng; fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits; NOTE: patients should stop using these fruits and herbal medications 7 days prior to first dose of study drug
* Primary central nervous system (CNS) lymphoma or active metastases to the CNS; NOTE: active is defined as requiring therapy such as surgery, radiation, or chemotherapy =< 28 days of study registration or ongoing corticosteroid therapy for CNS disease
* The following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * >= Common Terminology Criteria of Adverse Events (CTCAE) grade 3 anxiety
  * Meets the cut-off score of >= 12 in the Patient Health Questionnaire (PHQ)-9 or a cut-off of >= 15 in the Generalized Anxiety Disorder (GAD)-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to study registration; NOTE: erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to study registration, may be continued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Clinical benefit defined as a PR or CR as the objective status at any time or an objective status of SD for a duration of greater than 6 months from registration | From 6 months from registration up to 1 year
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent binomial confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Duration of response | From the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented, assessed up to 1 year
  If an adequate number of events are seen, the distribution of duration of response will be estimated using the method of Kaplan-Meier. Otherwise, duration of response will be summarized descriptively.
Overall response rate estimated by the number of confirmed responses (PR or CR) observed in the trial divided by the total number of evaluable patients | Up to 1 year
  Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Prognostic factors for aggressive lymphoma | Up to 1 year
  Will be summarized and used to help characterize the types of patients accrued to this trial. These classifications will be correlated with clinical benefit using Fisher's exact or Wilcoxon rank sum tests.
Progression-free survival time | Time from registration to progression or death due to any cause, assessed up to 1 year
  Will be estimated using the method of Kaplan-Meier.
Survival time | Time from registration to death due to any cause, assessed up to 1 year
  Will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Witzig, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States